CLINICAL TRIAL: NCT04921735
Title: An Observational Study of Cisatracurium 0.15 mg/kg, Comparing Onset Time, Duration of Action and Effect on Intubating Conditions in Young (18 - 40 Years) and Elderly (≥ 80 Years) Patients.
Brief Title: An Observational Study of Cisatracurium 0.15 mg/kg in Young and Elderly (≥ 80 Years) Patients.
Status: Completed | Type: Observational
Sponsor: Matias Vested (Other)
Responsible Party: Sponsor-Investigator, Matias Vested, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: Cisatracurium 2021
Record Dates: First submitted 2021-06-05; First posted 2021-06-10 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Onset Time of Cisatracurium; Duration of Action of Cisatracurium; Intubation Conditions
MeSH Terms: interventions — cisatracurium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elderly: patients aged 80 years or older
  Interventions: Drug: Cisatracurium
- young: patients aged 18-40 years
  Interventions: Drug: Cisatracurium

INTERVENTIONS:
Drug: Cisatracurium — 0.15 mg/kg based on ideal body weight calculated as height (cm) minus 105 for women and height (cm) minus 100 for men or actual body weight, whichever is lower

SUMMARY:
The aim of this study is to determine the onset time, duration of action and effect on intubation conditions of cisatracurium 0.15 mg/kg in elderly patients with age ≥ 80 years and in young patients aged 18 - 40 years.

DETAILED DESCRIPTION:
The aim of this study is to determine the onset time, duration of action and effect on intubation conditions of cisatracurium 0.15 mg/kg in elderly patients with age ≥ 80 years and in young patients aged 18 - 40 years. The hypothesis of this study is that cisatracurium administered in elderly patients (>80 years) has a longer onset time and duration of action compared to younger patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 80 or ≥18 - ≤40 years of age
2. Informed consent
3. Scheduled for elective surgery under general anaesthesia (expected duration of anaesthesia > 1 hour) with intubation and use of cisatracurium
4. American Society of Anaesthesiologists (ASA) physical status classification I to III
5. Can read and understand Danish

Exclusion Criteria:

1. Known allergy to cisatracurium
2. Neuromuscular disease
3. Indication for rapid sequence induction
4. Surgery in the prone position

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients (≥ 80 years) and younger patients (18-40 years) scheduled for elective surgery
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2021-12-19 (Actual)

PRIMARY OUTCOMES:
Onset time | within 10 minutes after administration
  the time from the start of the injection of cisatracurium to train-of-four (TOF) count of 0 monitored by acceleromyography

SECONDARY OUTCOMES:
Duration of action | within 120 minutes after administration of cisatracurium
  Duration of action is defined as time from start of cisatracurium injection to reappearance of TOF ratio > 0.9.
intubation conditions | within 10 minutes after administration of cistracurium
  intubation conditions are rated according to intubating difficulty score IDS when TOF-ratio is 0.
intubation conditions | within 10 minutes after administration of cisatracurium
  intubation conditions are rated according to Fuchs-Buder score when TOF-ratio is 0.
Laryngeal morbidity | 24 hours after surgery
  After 24 hours patients are asked about hoarseness and sore throat. Patients who experience either or both will be called 3 days postoperatively again. These two variables are assessed using a numeric ranking scale from 0 to 10.
Amount of ephedrine or metaoxedrine administered | within 10 minutes after administration of cisatracurium
  If ephedrine or metaoxedrine is administered after induction of anaesthesia and until the patient is ready for properly positioning for surgery, it will be noted in the CRF, as well as the amount administered. Changes in blood pressure or heart rate are treated according to local guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vested M, Kristensen CM, Pape P, Vang M, Hartoft M, Hjelmdal C, Rasmussen LS. Comparison of onset time, duration of action, and intubating conditions after cisatracurium 0.15 mg/kg in young and elderly patients. BMC Anesthesiol. 2022 Nov 7;22(1):339. doi: 10.1186/s12871-022-01881-5. PMID 36344924